CLINICAL TRIAL: NCT03649841
Title: Radiation Enhancement of Local and Systemic Anti-Prostate Cancer Immune Responses
Brief Title: Antiandrogen Therapy, Abiraterone Acetate, and Prednisone With or Without Neutron Radiation Therapy in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual.
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Zeng, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1001784; NCI-2018-01548 (Registry Identifier: NCI); 9938 (Other: FHCRC); P50CA097186 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Prostate Small Cell Neuroendocrine Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Abiraterone Acetate; Prednisone; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ADT, abiraterone, prednisone) (Active Comparator): Patients receive ADT per standard of care. Beginning 2 months after start of ADT, patients also receive abiraterone acetate and prednisone per standard of care for at least 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Antiandrogen Therapy; Drug: Abiraterone Acetate; Drug: Prednisone
- Arm II (ADT, abiraterone, prednisone, radiation therapy) (Experimental): Patients receive ADT, abiraterone acetate, and prednisone as in Arm I. Beginning 8-10 weeks after starting ADT and within 1 week of starting abiraterone acetate, patients also undergo 3-5 fractions of neutron radiation therapy for 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Antiandrogen Therapy; Drug: Abiraterone Acetate; Drug: Prednisone; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Antiandrogen Therapy — Undergo ADT
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Drug: Abiraterone Acetate — Undergo Abiraterone Acetate Treatment SOC
  Other Names: 17-(3-Pyridyl)-5,16-androstadien-3beta-acetate; 154229-18-2; Yonsa; Zytiga
Drug: Prednisone — Undergo Prednisone Treatment SOC
  Other Names: 10023; Delta 1-Cortisone
Radiation: Radiation Therapy — Undergo neutron radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; NOS; Radiotherapeutics; radiotherapy; RT; ENERGY TYPE
  Arms: Arm II (ADT, abiraterone, prednisone, radiation therapy)

SUMMARY:
This phase II trial studies how well antiandrogen therapy, abiraterone acetate, and prednisone with or without neutron radiation therapy work in treating patients with prostate cancer. Hormone therapy such as antiandrogen therapy may fight prostate cancer by blocking the production and interfering with the action of hormones. Abiraterone acetate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Neutron radiation therapy uses high energy neutrons to kill tumor cells and shrink tumors. It is not yet known whether antiandrogen therapy, abiraterone acetate, and prednisone with or without neutron radiation therapy may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ADT per standard of care. Beginning 2 months after start of ADT, patients also receive abiraterone acetate and prednisone per standard of care for at least 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive ADT, abiraterone acetate, and prednisone as in Arm I. Beginning 8-10 weeks after starting ADT and within 1 week of starting abiraterone acetate, patients also undergo 3-5 fractions of neutron radiation therapy for 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of prostate adenocarcinoma with < 50% neuroendocrine differentiation or small cell histology.
* At least one site of nodal or distant metastatic disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, or a bony metastasis that is evaluable on both computed tomography (CT) and bone scan.
* No prior orchiectomy.
* No androgen deprivation therapy such as treatment with antiandrogens, luteinizing hormone-releasing hormone (LHRH) agonists or antagonists for at least one year prior to trial enrollment, and testosterone must be inside normal range prior to trial enrollment if there is prior history of ADT.
* No other systemic anti-cancer therapy for at least 1-year prior to enrollment.
* Prior prostate-directed therapies such as prostatectomy or cryotherapy are allowed.
* Prior radiation treatments are allowed (prostate or metastatic sites) but must have been completed at least 3 months prior to starting ADT for this trial.
* White blood cell (WBC) > 3000/mm^3.
* Absolute neutrophil count (ANC) > 1000/mm^3.
* Platelets > 100,000/mm^3.
* Creatinine < 1.5 institutional upper limit of normal (ULN) or calculated creatinine clearance > 30 ml/min.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin < 3 x institutional ULN (unless patient has documented Gilbert's syndrome).
* No steroids for at least 2 weeks prior to enrollment, and patient must not be expected to require steroids during the study period, other than the typical low dose steroid that is given with abiraterone (typically prednisone or prednisolone at 5 mg twice daily).
* Zubrod performance status 0-2.
* Patient must sign study specific informed consent prior to study entry.
* Men who are sexually active must use medically acceptable forms of contraception.

Exclusion Criteria:

* Other illnesses with a life expectancy of less than 6 months, including but not limited to unstable angina, symptomatic congestive heart failure, cardiac arrhythmias.
* Psychological or social issues that would prevent patients from informed consent or complying with study requirements.
* Subject has a history of unexplained loss of consciousness or transient ischemic attack within 12 months of treatment start.
* Individuals on active treatment for a different cancer are excluded. Individuals with a history of other malignancies are eligible if they are deemed by the investigator to be at low risk for recurrence of that malignancy.
* Known brain metastasis.
* Known allergies, hypersensitivity, or intolerance to abiraterone or prednisone.
* Prior ADT less than a year, or greater than two months, prior to trial enrollment or prior ADT with testosterone less than normal.
* There is a potential drug interaction when abiraterone is concomitantly used with a CYP2D6 substrate narrow therapeutic index (e.g., thioridazine, dextromethorphan), or strong CYP3A4 inhibitors (e.g., atazanavir, erythromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole) or strong inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine). Caution should be used when patients are on one of these drugs.
* Patients with a history of pituitary or adrenal dysfunction, active or symptomatic viral hepatitis, human immunodeficiency virus (HIV), or chronic liver disease are not eligible.
* Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone once daily.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — University of Washington
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (ADT, Abiraterone, Prednisone) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy)
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (ADT, Abiraterone, Prednisone) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy) | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (6.1) | 64.3 (12) | 63.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Peripheral Blood Effector T-cells (CCR7-/CD45RO)
Description: Percent change in peripheral blood effector T-cells will be calculated by measuring the difference of the percent peripheral blood effector T-cells for each patient between two time points: pre-treatment and post-treatment (3 months after start of ADT, which is also 1 month post-radiation in the radiation arm). Unpaired two-sample t-test or Wilcoxon rank-sum test, depending on distribution of the percent change, will be used to test the null hypothesis that the percent change in peripheral blood effector T-cells is equal between the two arms.
Time Frame: Baseline to 3 months after start of antiandrogen therapy (ADT)
Population: Clinical trial closed early due to poor accrual. Enrolled patient numbers are much lower than expected (10 out of 30 patients enrolled). There is no funding to run the assays to analyze the data since the trial failed to complete accrual. The original collaborators who were supposed to pay for the assays withdrew due to low patient numbers, and lack of ability to draw scientific conclusions from low patient numbers.
Arm/Group | Arm I (ADT, Abiraterone, Prednisone) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rate of Undetectable Prostate Specific Antigen (PSA) (< 0.2)
Description: The number of patients with undetectable PSA at 6-months will be summarized by each arm and all combined.
Time Frame: At 6 months after start of abiraterone acetate
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (ADT, Abiraterone, Prednisone) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy)
Number analyzed (Participants) | 6 | 4
Participants | 1 | 1

3. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Safety and tolerability as evaluated by the incidence, severity, duration, causality, seriousness of adverse events. Toxicities will be summarized as the number of patients with grade 3 or higher toxicities per CTCAE v4.0, in addition to total number of toxicities (allowing for multiple toxicities within a patient) among all patients, and per treatment arm.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (ADT, Abiraterone, Prednisone) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy)
Number analyzed (Participants) | 6 | 4
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Start of Abiraterone to 6 months after start of Abiraterone. Total duration 6 months.
Description: Patients are seen in clinic every 4 weeks during the 6 months period above, and adverse events are scored per CTCAE v4.0 per physician reported outcomes.
Arm/Group | Arm I (ADT, Abiraterone, Prednisone) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (ADT, Abiraterone, Prednisone) (N=6) | Arm II (ADT, Abiraterone, Prednisone, Radiation Therapy) (N=4)
ALT elevation (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 2 ALT elevation
Headache (Nervous system disorders) | 1 (1) | NA — Grade 1 headaches

LIMITATIONS AND CAVEATS:
Early termination due to poor patient accrual leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03649841/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03649841/ICF_000.pdf